CLINICAL TRIAL: NCT05721586
Title: Effectiveness of Self-assembling Peptide (p11-4) in Conjunction With Fluoride Varnish in the Management of White Spot Lesions in Primary Teeth (Randomized Controlled Clinical Trial)
Brief Title: Self-assembling Peptide With Sodium Fluoride in Treating White Spot Lesionss in Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P11-4_2020
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: White Spot Lesion
MeSH Terms: interventions — Duraflor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CURODONTTM REPAIR: + Fluoride varnish (DURAFLOR) (Experimental)
  Interventions: Other: Self Assembling Peptide P11-4 (CURODONTTM REPAIR) + Fluoride varnish (DURAFLOR
- Fluoride Varnish (DURAFLOR) only (Active Comparator)
  Interventions: Other: Fluoride varnish (DURAFLOR

INTERVENTIONS:
Other: Self Assembling Peptide P11-4 (CURODONTTM REPAIR) + Fluoride varnish (DURAFLOR — The WSL was Acid etched with phosphoric acid gel 35-37% for 20 seconds, the tooth surface was rinsed with water and then dried afterwards application of CURODONTTM REPAIR
  Arms: CURODONTTM REPAIR: + Fluoride varnish (DURAFLOR)
Other: Fluoride varnish (DURAFLOR — A very thin coat of the DURAFLOR varnish was applied by a thin brush which was then allowed to dry for 10 seconds. The varnish hardens on contact with saliva or moisture
  Arms: Fluoride Varnish (DURAFLOR) only

SUMMARY:
Regenerative medicine-based approaches for caries treatment focus on biomimetic remineralization of initial carious lesions as a minimally invasive therapy using Self-Assembling Peptide P11-4 (CURODONTTM REPAIR) which enhances remineralization of white spot lesions (WSLs). The study aimed to assess clinically the effect of Self Assembling Peptide P11-4 (CURODONTTM REPAIR) + Fluoride varnish (DURAFLOR) versus a 5% fluoride varnish (DURAFLOR) on remineralization of enamel White Spot Lesions in primary teeth.

ELIGIBILITY:
Inclusion Criteria:

* children with high caries risk with the presence of at least one visible active WSL in primary teeth with ICDAS II score of 1, 2 or 3

Exclusion Criteria:

* Children with systemic diseases
* Teeth with cavitated lesion involving dentin and enamel defects

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Change in DIAGNOdent readings | Baseline, 3 months, and 6 months
  The measurements with the DIAGNOdent device that provides numerical values from 0 to 99

SECONDARY OUTCOMES:
Change in ICDAS II scores | Baseline, 3 months, and 6 months
  Code 0 Sound tooth surface:
  Code 1: First visual change in enamel. Code 2: Distinct visual change in enamel visible when wet, lesion must be visible when dry.
  Code 3: Localized enamel breakdown because of caries with no visible dentin or underlying shadow.
  Code 4: Underlying dark shadow from dentin with or without localized enamel breakdown.
  Code 5: Distinct cavity with visible dentin. Code 6: Extensive distinct cavity with visible dentin. After treatment, the evaluation will be performed as follows.
Change in Nyvad scores | Baseline, 3 months, and 6 months
  Code 0: Sound - Normal enamel
  Code 1: Active caries (intact surface) - Surface of enamel is whitish/yellowish opaque
  Code 2: Active caries (surface discontinuity)
  Code 3: Active caries (cavity) - Enamel/dentin cavity easily visible with the naked eye.
  Code 4: Inactive caries (intact surface) - Surface of enamel is whitish, brownish or black.
  Code 5: Inactive caries (surface discontinuity) - Same criteria as score 4. Localized surface defect (microcavity) in enamel only Code 6: Inactive caries (cavity) - Enamel/dentin cavity easily visible with the naked eye; surface of cavity may be shiny and feels hard on probing with gentle pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt